CLINICAL TRIAL: NCT04312945
Title: Affective Social Buffering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006378-2
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Social Stress; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary Parent (Experimental): Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, No Social Partner.
  In this case, the primary parent was present in the MRI room during the assessment.
  Interventions: Other: Questionnaires; Other: MRI
- Close Friend (Experimental): Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend,No Social Partner.
  In this case, the close friend was present in the MRI room during the assessment.
  Interventions: Other: Questionnaires; Other: MRI
- No Social Partner (Experimental): Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, No Social Partner.
  In this case, no social partner was present in the MRI room during the assessment.
  Interventions: Other: Questionnaires; Other: MRI

INTERVENTIONS:
Other: Questionnaires — The participant will complete questionnaires, including ones on pubertal development and quality of relations with parents and friends.
Other: MRI — Within 2 weeks of the first study visit, the participant will return to the University where they will undergo MRI.

SUMMARY:
The purpose of this experiment is to determine the mechanisms through which parental buffering of stress physiology during affective stimulus presentation diminishes with pubertal development and whether this diminution of effectiveness extends to social buffering by peers (best friends), in comparison to a lack of social partners.

DETAILED DESCRIPTION:
On visit one, the participant will complete questionnaires, including ones on pubertal development, screening for MRI safety, and quality of relations with parents and friends.

Within 2 weeks the participant will return to the University where they will undergo the following protocol. Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the scanner room: Primary Parent, Close Friend, No Social Partner. (N=50 per condition, 25 male, 25 female).

Once at the Center for Magnetic Resonance Research, participants and the individual who will be with the participant in the scanning room will undergo an MRI safety screening (the repeat of what was completed over the phone). Females will be shown to a changing room where the investigators will privately question them about any possibility of pregnancy. The participant will also have a chance to experience a simulated MRI in order to determine whether they will be comfortable in an actual MRI. Participants will be shown into the scanning control room and one more safety check will be performed before they enter the scanner room and the scanner. If they are in one of the social buffering conditions, the social buffering partner will also enter the scanning room and will sit to the side of the scanner.

The scanning bed will then be moved into the barrel of the MRI machine. The participant will be wearing head phones to protect his/her hearing and to receive instructions from the control room. The participant will then complete two emotionally evocative paradigms. The investigators will use a 3T Siemens Prisma scanner with a standard 32-channel phased array head coil.

ELIGIBILITY:
Inclusion Criteria:

* sufficient vision to complete assent and study procedures
* sufficient hearing to complete assent and study procedures
* sufficient language skills to provide verbal and written assent

Exclusion Criteria:

* Premature birth (less than 37 weeks)
* congenital and/or chromosomal disorders (e.g. cerebral palsy, FAS, mental retardation, Turner Syndrome, Down Syndrome, Fragile X)
* Autism Spectrum Disorders
* history of serious medical illness (e.g., cancer, organ transplant)
* youth taking systemic glucocorticoids
* youth taking beta-adrenergic medications
* diagnoses of psychiatric illness, seizure disorder or other neurological disorders
* contraindications for MRI (implanted medical device; presence of non-removal metal in or on the body, including piercings, orthodontic braces or certain permanent retainers)
* known pregnancy
* tattoos
* history of significant claustrophobia

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Gunnar, PhD, Principal Investigator — University of Minnesota; Kathleen Thomas, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Parent: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, No Social Partner.
  In this case, participants will complete the assessment with the primary parent in the MRI room.
- Close Friend: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend,No Social Partner.
  In this case, participants will complete the assessment with their close friend in the MRI room.
- No Social Partner: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, No Social Partner.
  In this case, participants will complete the assessment with no social partner in the MRI room.
Period: Overall Study
Arm/Group | Primary Parent | Close Friend | No Social Partner
Started | 69 | 69 | 64
Completed | 64 | 66 | 63
Not Completed | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- No Social Partner; Close Friend: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend,No Social Partner.
  Questionnaires: The participant will complete questionnaires, including ones on pubertal development and quality of relations with parents and friends.
  MRI: Within 2 weeks of the first study visit, the participant will return to the University where they will undergo MRI.
- Primary Parent: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, No Social Partner.
  Questionnaires: The participant will complete questionnaires, including ones on pubertal development and quality of relations with parents and friends.
  MRI: Within 2 weeks of the first study visit, the participant will return to the University where they will undergo MRI.
- Total: Total of all reporting groups
Arm/Group | No Social Partner | Primary Parent | Close Friend | Total
Number analyzed (Participants) | 63 | 64 | 66 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63 | 64 | 66 | 193
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 32 | 94
  Male | 33 | 32 | 34 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 54 | 51 | 55 | 160
  More than one race | 5 | 6 | 8 | 19
  Unknown or Not Reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 5 | 14
  Not Hispanic or Latino | 58 | 60 | 59 | 177
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cortisol AUCi
Description: Area under the curve from initial (baseline) will be calculated and used in the analyses. Description = 7 saliva samples are collected during the course of the assessment. These samples are collected at (1) arrival for training purposes, (2) scan preparation, (3) entering scanner, (4) pre-Hariri task, (5) post-Hariri, pre-IAPS GoNoGo task, (6) exiting scanner, (7) departure. Area under the curve at intercept (AUCi) is calculated using sample 2 as the intercept. This AUCi calculation samples 2 to 7, spanning approximately 100 minutes.
Time Frame: 2 hours
Population: 193 participants were completed, with 63 Alone, 64 Parent, and 66 Friend. For each outcome, all available analyzable data were included in results, sometimes resulting in lower n.
Measure: Mean (Standard Deviation); unit: (ug/dL)*minutes
Groups:
- No Social Partner: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend,No Social Partner.
  In this case, no social partner was present in the MRI room during the assessment.
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 57 | 56 | 54
(ug/dL)*minutes | -93.6397 (182.94398) | -68.0959 (239.64667) | -106.9105 (227.39856)

2. Primary Outcome: Change Heart Rate Response
Description: Heart rate will be derived from the pulse-oximeter signal collected during periods of emotional affect and rest during the course of the assessment. The variable, heart rate response, is a numeric output (beats per minute) from validated software (BIOPAC). The outcome measure will be reported (in beats per minute) as the difference between heart rate response during the period of emotional affect and period of rest.
Time Frame: period of resting state fMRI and period of emotional task fMRI (approximately 5 minutes after rest)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Primary Parent: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend, No Social Partner.
- Close Friend; No Social Partner: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend,No Social Partner.
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 26 | 28 | 32
beats per minute | .543 (3.818) | .707 (2.418) | 1.343 (3.106)

3. Primary Outcome: Left Amygdala: Task-related Brain Activity During Hariri Task
Description: The change in fMRI signal intensity in the left amygdala between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
% change in BOLD signal | 0.231 (0.136) | 0.245 (0.153) | 0.232 (0.151)

4. Primary Outcome: Left Amygdala: Task-related Brain Activity During IAPS GoNoGo Task
Description: The difference in fMRI signal intensity in the left amygdala between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 51 | 56
% change in BOLD signal | 0.28073 (.15741) | .29334 (.18174) | .29397 (.15677)

5. Primary Outcome: Right Amygdala: Task-related Brain Activity During Hariri Task
Description: The change in fMRI signal intensity in the right amygdala between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
% change in BOLD signal | 0.275 (0.140) | 0.273 (0.164) | 0.297 (0.151)

6. Primary Outcome: Right Amygdala: Task-related Brain Activity During IAPS GoNoGoTask
Description: The difference in fMRI signal intensity in the right amygdala between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 51 | 56
% change in BOLD signal | 0.30121 (0.19301) | 0.29021 (0.18815) | 0.33038 (0.15398)

7. Primary Outcome: Left Insula: Task-related Brain Activity During Hariri Task
Description: The change in fMRI signal intensity in the left insula between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
% change in BOLD signal | -0.008 (0.124) | 0.0007 (0.153) | -0.018 (0.129)

8. Primary Outcome: Left Insula: Task-related Brain Activity During IAPS GoNoGo Task
Description: The difference in fMRI signal intensity in the left insula between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 51 | 56
% change in BOLD signal | .01627 (.14347) | .02078 (.15591) | .00809 (.15488)

9. Primary Outcome: Right Insula: Task-related Brain Activity During Hariri Task
Description: The change in fMRI signal intensity in the right insula between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
% change in BOLD signal | -0.012 (0.136) | 0.0004 (0.144) | -0.017 (0.100)

10. Primary Outcome: Right Insula: Task-related Brain Activity During IAPS GoNoGo Task
Description: The difference in fMRI signal intensity in the right insula between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 51 | 56
% change in BOLD signal | .01504 (.14045) | .01356 (.18215) | -0.00077 (.12285)

11. Primary Outcome: Dorsomedial Prefrontal Cortex (dmPFC): Task-related Brain Activity During Hariri Task
Description: The change in fMRI signal intensity in the bilateral dorsomedial prefrontal cortex (dmPFC) between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
% change in BOLD signal | 0.048 (0.190) | 0.093 (0.218) | 0.108 (0.227)

12. Primary Outcome: Dorsomedial Prefrontal Cortex (dmPFC): Task-related Brain Activity During IAPS GoNoGo Task
Description: The difference in fMRI signal intensity in the bilateral dorsomedial prefrontal cortex (dmPFC) between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in BOLD signal
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 51 | 56
% change in BOLD signal | .02224 (.20273) | .02385 (.20474) | .00827 (.17163)

13. Primary Outcome: Amygdala-vmPFC: Psychophysiological Interaction (PPI) Functional Connectivity During Hariri Task
Description: For each participant, blood oxygenation level dependent (BOLD) signal intensity (unitless measure) will be measured using fMRI in the bilateral amygdala over a five-minute recording period. Signal intensity will also be measured using fMRI in the ventromedial prefrontal cortex (vmPFC) over the same period of time. An interaction analysis will be conducted to measure the effect of task condition on bilateral amygdala-vmPFC functional connectivity, which will be reported as a Z-score. A Z-score of zero indicates no difference in amygdala-vmPFC functional connectivity as a function of task. A more positive Z-score indicates increased amygdala-vmPFC functional connectivity during the emotional blocks of the task relative to the control blocks. A more negative Z-score indicates decreased amygdala-vmPFC functional connectivity during the emotional blocks of the task relative to the control blocks.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
Z-score | -0.033 (0.453) | -0.033 (0.428) | 0.116 (0.445)

14. Primary Outcome: Amygdala-vmPFC: Psychophysiological Interaction (PPI) Functional Connectivity During IAPS GoNoGo Task
Description: For each participant, blood oxygenation level dependent (BOLD) signal intensity (unitless measure) will be measured using fMRI in the bilateral amygdala over a ten-minute recording period. Signal intensity will also be measured using fMRI in the ventromedial prefrontal cortex (vmPFC) over the same period of time. An interaction analysis will be conducted to measure the effect of task condition on bilateral amygdala-vmPFC functional connectivity, which will be reported as a Z-score. A Z-score of zero indicates no difference in amygdala-vmPFC functional connectivity as a function of task. A more positive Z-score indicates increased amygdala-vmPFC functional connectivity during the emotional blocks of the task relative to the control blocks. A more negative Z-score indicates decreased amygdala-vmPFC functional connectivity during the emotional blocks of the task relative to the control blocks.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 50 | 56
Z-score | -0.11810 (.54062) | .01399 (.53853) | -0.01128 (.49507)

15. Primary Outcome: Amygdala-dmPFC: Psychophysiological Interaction (PPI) Functional Connectivity During Hariri Task
Description: For each participant, blood oxygenation level dependent (BOLD) signal intensity (unitless measure) will be measured using fMRI in the bilateral amygdala over a five-minute recording period. Signal intensity will also be measured using fMRI in the dorsomedial prefrontal cortex (dmPFC) over the same period of time. An interaction analysis will be conducted to measure the effect of task condition on bilateral amygdala-dmPFC functional connectivity, which will be reported as a Z-score. A Z-score of zero indicates no difference in amygdala-dmPFC functional connectivity as a function of task. A more positive Z-score indicates increased amygdala-dmPFC functional connectivity during the emotional blocks of the task relative to the control blocks. A more negative Z-score indicates decreased amygdala-dmPFC functional connectivity during the emotional blocks of the task relative to the control blocks.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 56 | 53 | 55
Z-score | 0.055 (0.326) | 0.127 (0.321) | 0.072 (0.393)

16. Primary Outcome: Amygdala-dmPFC: Psychophysiological Interaction (PPI) Functional Connectivity During IAPS GoNoGo Task
Description: For each participant, blood oxygenation level dependent (BOLD) signal intensity (unitless measure) will be measured using fMRI in the bilateral amygdala over a ten-minute recording period. Signal intensity will also be measured using fMRI in the dorsomedial prefrontal cortex (dmPFC) over the same period of time. An interaction analysis will be conducted to measure the effect of task condition on bilateral amygdala-dmPFC functional connectivity, which will be reported as a Z-score. A Z-score of zero indicates no difference in amygdala-dmPFC functional connectivity as a function of task. A more positive Z-score indicates increased amygdala-dmPFC functional connectivity during the emotional blocks of the task relative to the control blocks. A more negative Z-score indicates decreased amygdala-dmPFC functional connectivity during the emotional blocks of the task relative to the control blocks.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 54 | 50 | 56
Z-score | .01220 (.43335) | .008081 (.30828) | .04997 (.37726)

17. Primary Outcome: Change in EDA During Hariri Task
Description: The difference in mean amplitude EDA response between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microSiemens
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 25 | 22 | 23
microSiemens | .001569 (.0221798) | .000659 (.0089826) | -0.01369 (.0190926)

18. Primary Outcome: Change in EDA During IAPS GoNoGo Task
Description: The difference in mean amplitude EDA response between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microSiemens
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 24 | 23 | 33
microSiemens | .002348 (.0208932) | .003808 (.0106093) | .000465 (.0141820)

19. Primary Outcome: EDA at Rest
Description: EDA response amplitude during rest.
Time Frame: during resting state fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microSiemens
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 28 | 26 | 31
microSiemens | .0269 (.01828) | .0273 (.01586) | .0287 (.02013)

20. Secondary Outcome: Change in Self Report of Stress
Description: The Self Report of Stress is an 8-item questionnaire assessing participant level of stress at various time points across the session. Items are rated on a 5 point Likert scale. Total score is the unweighted mean of item scores. Total scores range from 0 to 40, with higher scores indicating greater stress. The assessment will be administered at baseline (no stress) and during a period of stress. The outcome will be reported as the difference between the baseline period and experimental stress period.
Time Frame: start of 2 hr testing session and period of emotional affect tasks (approx. 105 minutes after start)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 60 | 60 | 59
scores on a scale | 0.0000 (.4500) | .4500 (1.20978) | .3305 (1.0692)

21. Secondary Outcome: Change in Accuracy During Hariri Task
Description: Change in accuracy for stimulus matching between the emotional and non-emotional stimuli during the task.
Time Frame: during Hariri task fMRI scan (approx. 5 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in accuracy
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 60 | 60 | 59
% change in accuracy | -25.27 (16.717) | -25.37 (24.261) | -25.31 (19.498)

22. Secondary Outcome: Change in Accuracy During IAPS GoNoGo Task
Description: Change in accuracy of go/no go (press for go trials and no-press for no go trials) between the negative affect and scrambled stimuli during the task.
Time Frame: during GoNoGo task fMRI scan (approx. 10 minute duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in accuracy
Arm/Group | Primary Parent | Close Friend | No Social Partner
Number analyzed (Participants) | 59 | 59 | 58
% change in accuracy | -2.01 (6.129) | -0.86 (6.311) | -2.50 (5.269)

ADVERSE EVENTS:
Time Frame: during testing session, 2 hours
Groups:
- No Social Partner: Participants will be randomly assigned to one of 3 conditions that differ by who is with them in the MRI scanner room: Primary Parent, Close Friend,No Social Partner.
  In this case, the no social partner was present in the MRI room during the assessment.
Arm/Group | Primary Parent | Close Friend | No Social Partner
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/66 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04312945/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04312945/ICF_001.pdf